CLINICAL TRIAL: NCT01084785
Title: Storing Blood for Analysis of DNA and Protein of Patients With Cancer in MAASTRO Clinic
Brief Title: Biobank Carcinoma: Storing Blood and Protein of Patients With Cancer
Acronym: Biobank
Status: Recruiting | Type: Observational
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 08-06-23/01; NCT00157352 (obsolete NCT alias); NCT00157365 (obsolete NCT alias); NCT00157391 (obsolete NCT alias); NCT00157404 (obsolete NCT alias); NCT00157417 (obsolete NCT alias); NCT00157430 (obsolete NCT alias); NCT00157443 (obsolete NCT alias); NCT00157456 (obsolete NCT alias); NCT00157469 (obsolete NCT alias); NCT00157495 (obsolete NCT alias); NCT00181337 (obsolete NCT alias); NCT00181376 (obsolete NCT alias); NCT00181389 (obsolete NCT alias); NCT00181402 (obsolete NCT alias); NCT00181415 (obsolete NCT alias); NCT00181428 (obsolete NCT alias); NCT00181441 (obsolete NCT alias); NCT00181454 (obsolete NCT alias); NCT00181467 (obsolete NCT alias); NCT00181480 (obsolete NCT alias); NCT00181493 (obsolete NCT alias); NCT00181519 (obsolete NCT alias); NCT01067872 (obsolete NCT alias)
Record Dates: First submitted 2010-03-10; First posted 2010-03-11 (Estimated); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Cancer
Keywords: Cancer; genomics; proteomics
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine, by means of DNA and protein analysis, the relationship between DNA and protein profiles and a number of endpoints, which are important for the patient such as overall survival and side effects.

DETAILED DESCRIPTION:
It has already been known for a long time that cancer is a genetic disorder and that the development of the illness is a very complex interaction between genetic and surrounding factors. Also the response on therapy and the development and seriousness of side effects is stipulated by this complicated collaboration of genetic and surrounding factors. Moreover it is not only the DNA that plays an important role but also the systems of control at protein level. At this moment a lot of questions remain to be answered because up till now the studies were of rather restricted statistic strength with frequently inconsistent dates and moreover retrospective. Major retrospective studies are necessary to distinguish the relationship between DNA/protein patterns and clinical relevant endpoints like prognosis and toxicity in which an as broad as possible patient group is being monitored. For this reason we want to take blood samples in MAASTRO clinic of all patients with lung cancer and to store it encrypted so that we can perform DNA and protein analyses in future and to correlate the results with survival and toxicity of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* cancer

Exclusion Criteria:

* not able to comply with follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2003-01-01; Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Dirk De Ruysscher, Prof PHD, Principal Investigator — CCMO
Locations (1):
- Maastricht Radiation Oncology, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Dehing-Oberije C, Aerts H, Yu S, De Ruysscher D, Menheere P, Hilvo M, van der Weide H, Rao B, Lambin P. Development and validation of a prognostic model using blood biomarker information for prediction of survival of non-small-cell lung cancer patients treated with combined chemotherapy and radiation or radiotherapy alone (NCT00181519, NCT00573040, and NCT00572325). Int J Radiat Oncol Biol Phys. 2011 Oct 1;81(2):360-8. doi: 10.1016/j.ijrobp.2010.06.011. Epub 2010 Oct 1. PMID 20888135